CLINICAL TRIAL: NCT01234285
Title: Safety of Heparin Anticoagulation for Prevention of Death in Patients With Septic Shock.
Brief Title: Safety of Heparin in Patients With Septic Shock
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sara Cheng, MD has left the Univ. of Colorado and the study has been closed.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0595
Record Dates: First submitted 2010-09-23; First posted 2010-11-04 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Sepsis
Keywords: sepsis; septic shock; anticoagulation; intensive care unit
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- intravenous heparin aPTT 40-50 seconds (Experimental): Patients 11-15: IV heparin, target aPTT range 40-50 seconds
  Interventions: Drug: heparin
- intravenous heparin (Experimental): Patients 26-40: IV heparin, target range aPTT 50-60 seconds
  Interventions: Drug: heparin
- Intravenous heparin (Experimental): Patients 41-55 IV heparin, target aPTT range 60-70 seconds
  Interventions: Drug: heparin
- sq heparin three times a day (Active Comparator): Patients 1-10 will receive subcutaneous heparin three times a day
  Interventions: Drug: heparin

INTERVENTIONS:
Drug: heparin — intravenous heparin titrated to an aPTT of 40-50 seconds starting between 300-500 units per hour and adjusted every 6 hours based on aPTT, starting within 24 hours of ICU admission up to 6 days.
  Arms: intravenous heparin aPTT 40-50 seconds
Drug: heparin — intravenous heparin titrated to an aPTT of 50-60 seconds starting between 300-500 units per hour and adjusted every 6 hours based on aPTT, starting within 24 hours of ICU admission up to 6 days.
  Arms: Intravenous heparin; intravenous heparin
Drug: heparin — intravenous heparin titrated to an aPTT of 40-45 seconds starting between 300-500 units per hour and adjusted every 6 hours based on aPTT, starting within 24 hours of ICU admission up to 6 days.
  Arms: Intravenous heparin; intravenous heparin
Drug: heparin — 5000 units subcutaneously three times a day, starting within 24 hours of ICU admission up to 6 days.
  Arms: sq heparin three times a day

SUMMARY:
Sepsis is a syndrome comprised of a systemic inflammatory response, signs of tissue hypoperfusion, and organ in the setting of presumed infection. Heparin, in addition to being an anticoagulant, is also a well-known antiinflammatory. The investigators believe that unfractionated heparin has the potential to save the lives of septic patients at a drastically reduced cost. This is a dose escalation study to determine the safety of increasing levels of heparin in this patient population; compare markers of anticoagulation and inflammation between treatment groups; and compare clinical outcomes between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-90 in the medical or surgical intensive care unit
2. Within 24 hours of diagnosis with sepsis as defined by the Bone criteria (see Appendix A);
3. Acute Physiology and Chronic Health Evaluation (APACHE II) score of > 25;
4. Signed consent

Exclusion Criteria:

1. Currently therapeutically anticoagulated for known thrombotic diagnosis (myocardial infarction, venous thromboembolism) known molecular hypercoagulable state (Factor V Leiden, lupus anticoagulant, antiphospholipid antibody syndrome); or use of cardiopulmonary support machines (left-ventricular assist device, intra-aortic balloon pump, veno-venous ultrafiltration, or extracorporeal membrane oxygenation.
2. History of gastrointestinal or cerebral hemorrhage within past 3 months;
3. Active bleeding;
4. Known allergy or sensitivity to heparin;
5. History of heparin-induced thrombocytopenia
6. Organ transplantation recipient -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of major bleeding | This outcome will be measured for an average of 30 days
  Defined as:decrease in hemoglobin greater than 2g/dl and/or transfusion of 2 or more units of packed red blood cells.
  However, if there are obvious other reasons for bleeding, such as within 12 hours of major surgery, coagulopathy unrelated to heparin or an anatomical basis.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cheng, MD;PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Marshall JC. Inflammation, coagulopathy, and the pathogenesis of multiple organ dysfunction syndrome. Crit Care Med. 2001 Jul;29(7 Suppl):S99-106. doi: 10.1097/00003246-200107001-00032. PMID 11445742
- [Background] Agarwal R, Gupta D. Anticoagulation in sepsis: is low-dose heparin as effective as activated protein C? Intensive Care Med. 2005 Sep;31(9):1297-8. doi: 10.1007/s00134-005-2723-0. Epub 2005 Jul 9. No abstract available. PMID 16007415
- [Background] Zarychanski R, Doucette S, Fergusson D, Roberts D, Houston DS, Sharma S, Gulati H, Kumar A. Early intravenous unfractionated heparin and mortality in septic shock. Crit Care Med. 2008 Nov;36(11):2973-9. doi: 10.1097/CCM.0b013e31818b8c6b. PMID 18824906
- [Background] Robertson MS. Heparin: the cheap alternative for immunomodulation in sepsis? Crit Care Resusc. 2006 Sep;8(3):235-8. PMID 16930112
- [Background] Derhaschnig U, Pernerstorfer T, Knechtelsdorfer M, Hollenstein U, Panzer S, Jilma B. Evaluation of antiinflammatory and antiadhesive effects of heparins in human endotoxemia. Crit Care Med. 2003 Apr;31(4):1108-12. doi: 10.1097/01.CCM.0000059441.70680.DC. PMID 12682480